CLINICAL TRIAL: NCT00465530
Title: Safety and Efficacy of Once Daily Intranasal Gentamycin Irrigation Versus Saline in the Treatment of Pediatric Chronic Sinusitis
Brief Title: Comparing the Use of Saline or Saline Plus Gentamycin in Nasal Irrigation to Treat Chronic Sinusitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Wei, MD (Other)
Responsible Party: Sponsor-Investigator, Julie Wei, MD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10553
Record Dates: First submitted 2007-04-23; First posted 2007-04-25 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-04

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Sodium Chloride; Gentamicins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): Saline plus Gentamycin
  Interventions: Drug: Saline; Drug: Gentamycin
- 1 (Placebo Comparator): Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — Intranasal Saline
Drug: Gentamycin — Intranasal irrigation
  Arms: 2

SUMMARY:
Healthy children may develop symptoms of chronic sinusitis such as chronic cough, chronic runny nose, nasal congestion, even headaches. Such symptoms may persist long after the child gets over other symptoms of a cold and commonly result in the prescription of oral antibiotics. The purpose of this study is to evaluate whether using saline alone or saline plus an antibiotic (gentamycin) to irrigate the nose directly once a day for 6 weeks is effective and safe for the treatment of the above named symptoms. Computerized axial tomography (CAT) scans and quality of life surveys will be used to compare the health of the sinuses before and after treatment, and scored to determine which of the two treatments, saline alone or saline with gentamycin, is more effective in the treatment of this condition. The study hypothesis is that intranasal saline irrigation will work as well as saline plus gentamycin, and that majority of the patients will experience significant improvement after a 6 week treatment period.

DETAILED DESCRIPTION:
In the pediatric population, rhinosinusitis is a common concern resulting frequently in the frequent and unsuccessful prescription of systemic oral antibiotic therapy. Children typically experience an estimated 6-8 upper respiratory illnesses per year, usually viral, and only 13% are estimated to result in true sinusitis. True and chronic sinusitis, if not adequately treated, may result in long term symptoms including nasal airway obstruction, nasal congestion, persistent mucopurulent rhinorrhea, daytime and nocturnal cough, headaches, daytime fatigue, and even exacerbation or poor control of underlying asthma. A child's quality of life can be severely impacted as is their caretaker's due to days of missed school, frequency of doctor visits and courses of oral antibiotic therapy prescribed for the above mentioned symptoms, which ultimately result in the development of resistant organisms in addition to potential negative side effects associated with systemic oral antibiotic use.

Intranasal saline irrigation is underutilized in the pediatric population, most likely due to the presumption that children will not cooperate nor tolerate the act of irrigation. Saline irrigation of the nose is an inexpensive and generally well tolerated treatment with very little side effects or risks. Rigorous data regarding the efficacy of saline irrigation has become more available in this past decade, with most studies demonstrating a clear improvement in patient quality of life as measured by various study instruments or outcome surveys.

In our protocol, patients will be randomized to receive either saline alone or saline plus gentamycin in the solution form for nasal irrigation once daily for a six week treatment period. Weekly phone calls will be made to check for possible adverse events while patients are on treatment, and at the end of the treatment period another CAT scan will be performed to assess the status of the sinuses. Overall improvement will be determined based on the sinus status on the second CAT scan as well as the quality of life survey filled out by parents.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children age 4-17
* History of "Recurrent" or "Chronic Sinusitis"

  * Definition: History must include > 3 months of any or a combination of the following symptoms:
  * Nasal congestion/nasal airway obstruction
  * Rhinorrhea/Nasal discharge
  * Persistent cough (daytime)
  * Postnasal drip
  * Headache
  * Facial pain
  * Foul breath
  * Intermittent fever
* Caregiver (proxy responsible) able to read and understand English
* Has had at least 3 courses or a total of 21 days of oral antibiotic therapy for above symptoms in the previous 3 months
* Child has a CT scan of the coronal sinus without contrast within two months prior to visit date, which demonstrates and opacification of a single or multiple, ipsilateral or bilateral sinuses.

Exclusion Criteria:

* Inability of caregiver to read and understand English
* Mental retardation, cognitive impairment, or developmental delay
* History of cystic fibrosis
* History of immotile cilia syndrome
* History of immune suppression/immune compromise
* CT scan within past 4 weeks available for review at time of clinic visit which is entirely negative for evidence of sinus disease plus complete absence of any of the above symptoms
* History of endoscopic sinus surgery
* History of patient's inability to tolerate attempted nasal irrigation in the past 6 months
* History of recent use of gentamycin intranasal irrigation or saline irrigation within the past 3 months
* History of presence of nasal polyposis
* History of allergic reaction of any kind to intravenous gentamycin or aminoglycosides in past medical history (for treatment of any infections)

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Wei, M.D., Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kansas MedWest, Shawnee, Kansas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline Plus Gentamycin (Once Daily, 40 mL to Each Nostril) | Saline (Once Daily, 40 mL to Each Nostril)
Started | 21 | 19
Completed | 19 | 15
Not Completed | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Plus Gentamycin (Once Daily, 40 mL to Each Nostril) | Saline (Once Daily, 40 mL to Each Nostril) | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 19 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 9 | 16 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change in Computed Tomography (CT) Score After Treatment
Description: Change in CT score reflects the Lund-Mackay staging system. Each sinus is scored separately and scores are determined for the right and the left side. The lowest score of 0 represents no opacification in the sinus. A score of 1 represents a partial opacification. A score of 2 represents complete opacification.
Time Frame: Change from Baseline to 6 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline (Once Daily, 40 mL to Each Nostril) | Saline Plus Gentamicin (Once Daily, 40 mL to Each Nostril)
Number analyzed (Participants) | 15 | 19
units on a scale
  Left maxillary | -.64 (.63) | -.63 (.5)
  Right maxillary | -.5 (.65) | -.5 (.63)
  Left anterior ethmoid | -.79 (.7) | -1.06 (.68)
  Right anterior ethmoid | -.79 (.8) | -.63 (.81)
  Left posterior ethmoid | -.57 (.65) | -.81 (.66)
  Right posterior ethmoid | -.64 (.63) | -.75 (.68)
  Left sphenoid | -.43 (.65) | -.5 (.73)
  Right sphenoid | -.5 (.65) | -.5 (.73)
  Left frontal | -.89 (.78) | -.56 (.53)
  Right frontal | -.8 (.63) | -.22 (.44)
  Left OMC | -1 (1.03) | -1.25 (1)
  Right OMC | -.86 (1.29) | -.88 (1.02)
  Total Score, left | -4.07 (3.25) | -4.56 (2.42)
  Total score, right | -3.86 (3.11) | -3.38 (2.66)

2. Secondary Outcome: Change in Overall Quality of Life
Description: Measured by Quality of Life Survey (SN-5). Scores ranged from 0 - 7. The higher the numerical score, the worse the problem.
Time Frame: Baseline to 3 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline (Once Daily, 40 mL to Each Nostril) | Saline Plus Gentamicin (Once Daily, 40 mL to Each Nostril)
Number analyzed (Participants) | 15 | 19
units on a scale | 2.53 (1.99) | 2.06 (2.88)

3. Primary Outcome: Change in Overall Quality of Life
Description: as for outcome 2
Time Frame: 3 Weeks to Follow-Up (7 Weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Saline (Once Daily, 40 mL to Each Nostril) | Saline Plus Gentamicin (Once Daily, 40 mL to Each Nostril)
Number analyzed (Participants) | 15 | 19
units on a scale | .69 (1.75) | 1.38 (1.75)

ADVERSE EVENTS:
Arm/Group | Saline Plus Gentamycin (Once Daily, 40 mL to Each Nostril) | Saline (Once Daily, 40 mL to Each Nostril)
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 3/21 | 6/19
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline Plus Gentamycin (Once Daily, 40 mL to Each Nostril) (N=21) | Saline (Once Daily, 40 mL to Each Nostril) (N=19)
Otalgia (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Symptoms of Allergic rhinitis (General disorders) | 1 (1) | 1 (1)
Acute otitis media (AOM) (General disorders) | 0 (0) | 2 (2)
Epistaxis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cough (General disorders) | 1 (1) | 0 (0)
Poison Ivy (General disorders) | 0 (0) | 1 (1)
Auditory (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes